CLINICAL TRIAL: NCT04316494
Title: Hydroxychloroquine in ANCA Vasculitis Evaluation - A Multicentre, Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Hydroxychloroquine in ANCA Vasculitis Evaluation
Acronym: HAVEN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 251987; 2018-001268-40 (EudraCT Number)
Record Dates: First submitted 2020-02-25; First posted 2020-03-20 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2023-08

CONDITIONS: ANCA Associated Vasculitis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Wegener Granulomatosis
Keywords: Granulomatosis Polyangiitis; Eosinophilic Granulomatosis with Polyangiitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Granulomatosis with Polyangiitis | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Central trial pharmacist will be unblinded during trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): Patients will be receive 400mg of Hydroxychloroquine (2 x 200mg) to take daily for 52 weeks. Hydroxychloroquine will be started at a dose of 200mg an up-titrated after the first week to a maximum daily dose of 400mg.
  Patients weighing <50kg, or those patients with an eGFR of 30-50mL/min, will receive a reduced dose of 200mg daily.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Patients will be receive 400mg of Placebo (2 x 200mg) to take daily for 52 weeks. Placebo will be started at a dose of 200mg an up-titrated after the first week to a maximum daily dose of 400mg.
  Patients weighing <50kg, or those patients with an eGFR of 30-50mL/min, will receive a reduced dose of 200mg daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — White, round, film-coated tablets marked 'HCQ' on one side and 200' on the other side.
  Excipients:
  Lactose monohydrate Maize Starch Magnesium Stearate Polyvidone Opadry OY-L-28900
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo — Placebo to match Hydroxychloroquine.
  Excipients:
  Microcrystalline cellulose Lactose Magnesium Stearate
  Other Names: Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out whether hydroxychloroquine, in addition to background treatments, reduces disease activity in patients with Anti-Neutrophilic Cytoplasmic Autoantibodies (ANCA) Vasculitis, a group of autoimmune diseases.

Hydroxychloroquine and is an established, effective, safe and inexpensive therapy, widely used in other autoimmune diseases such as lupus and rheumatoid arthritis.

The study is open to adults diagnosed with certain types of vasculitis, called Granulomatosis Polyangiitis (GPA), Microscopic Polyangiitis (MPA) or Eosinophilic Granulomatosis with Polyangiitis (EGPA). Participants will be eligible if they are treated with background medication to control their vasculitis disease and have a low level of disease activity as defined by a Birmingham Vasculitis Activity Score (BVAS) of greater than 3.

Participants will be randomly placed in 1 of 2 groups. Both groups will be given background medication. One group will receive hydroxychloroquine and the other will receive placebo. Participants will be on treatment for 1 year.

76 ANCA Vasculitis participants will be recruited (38 in each treatment arm) from UK vasculitis specialist centres.

DETAILED DESCRIPTION:
This is a multi-centre, randomised, placebo-controlled, double-blind study to evaluate if hydroxychloroquine in combination with background maintenance therapy improves the clinical response and quality of life in patients with AAV. 76 participants who have Granulomatosis with Polyangiitis, Microscopic Polyangiitis or Eosinophilic Granulomatosis with Polyangiitis will be recruited from 20 sites.

They will be randomised in a 1:1 ratio of hydroxychloroquine or placebo. Neither the patient nor the research team will know which treatment group the participant is in.

Once the participant agrees to take part and has signed informed consent, they will undergo the following assessments, tests and procedures to find out if they can take part in the study. Some may be routinely done by the study doctor as part of regular vasculitis care even if the participants are not in the study:

* Medical history
* Birmingham Vasculitis Activity Score (BVAS)
* Physical exam
* Blood tests
* Pregnancy test
* Urine drug test
* Electrocardiogram

If the patient is eligible to take part in the study, they will be randomised to receive either hydroxychloroquine or placebo in addition to background medication. Participants will receive 2 tablets to take once a day over the course of a year. Participants may have their dose reduced to 1 tablet dependent on their weight at baseline and renal function. All participants will have their prednisolone dose tapered down over the course of the study. Participants will be asked to fill in a patient diary on a weekly basis to record whether they've taken their medication, and if they've experienced any change of symptoms.

Participants will be asked to attend the hospital at weeks 4, 16, 28, 40, 44, 48, 52 and 56. At each of these visits, participants will undertake some or all of the following tests/assessments:

* Physical exam including visual acuity
* Weight and vital signs
* BVAS assessment and Vasculitis Damage Index (VDI)
* Patient questionnaires
* If there are any changes to their medicines and health status
* If they experiencing any side effects
* Blood samples and urine tests to see how the study drug is affecting the body.
* At two visits, participants will also be asked to undergo an electrocardiogram (ECG).

Patients will be followed up by phone in weeks 10, 22, and 34. This phone call will be based on the ANCA-associated Vasculitis Patient Reported Outcome (AAV PRO) questionnaire and patients will also be encouraged to report any adverse events. Patients reporting new or worsening symptoms will be invited to the hospital for an unscheduled visit.

In addition to clinical bloods, 76ml of blood will be taken for research purposes for all participants. These will be taken at the same time as clinical bloods to minimise discomfort for the participant. Participants at Guy's and St Thomas' will have an additional 200ml of blood taken for isolation of cells. These bloods will be stored and kept for future research, with the written consent of the participant.

ELIGIBILITY:
Inclusion Criteria

1. Are at least 18 years of age at screening.
2. Have a clinical diagnosis of Granulomatosis Polyangiitis (GPA) or a diagnosis of Microscopic Polyangiitis (MPA) or a diagnosis of Eosinophilic Granulomatosis with Polyangiitis (EGPA) according to the Chapel Hill criteria.
3. Have a Birmingham Vasculitis Activity Score >3 BVAS v.3 (Appendix 2) with minor BVAS items only (no major BVAS items).BVAS should be >3 at screening and at randomisation.
4. Patients should be receiving maintenance therapy at a stable dose for 4 weeks prior to randomisation. Maintenance therapy is defined as prednisolone and/or azathioprine, methotrexate, mycophenolate, co-trimoxazole or maintenance rituximab therapy.
5. Patients receiving corticosteroids for reasons other than vasculitis must be on a stable regimen for four weeks prior to randomisation.
6. A female patient is eligible to enter the study if she is:

   Not pregnant or nursing; OR Of non-childbearing potential (i.e., women who have had a hysterectomy, are postmenopausal defined as ≥1 year without menses, have both ovaries surgically removed or have documented tubal ligation or other permanent sterilization procedure); OR

   Of childbearing potential. These women must have a negative urine pregnancy test at screening and at baseline and be using at least one effective method of contraception. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Consistent and correct use of one of the following acceptable methods of birth control for 1 month prior to the start of the study agent, during the study, and 16 weeks after the last dose of study agent:

   Oral contraceptive, either combined or progestogen alone Injectable progestogen Implants of levonorgestrel or etonogestrel Estrogenic vaginal ring Percutaneous contraceptive patches Intrauterine device (IUD) or intrauterine system (IUS) with <1% failure rate as stated in the product label
7. No contraindications to hydroxychloroquine therapy.
8. Willing and able to give written informed consent to participate in the trial.
9. Patients should have sufficient English in order to provide informed consent and complete the patient questionnaires.

Exclusion Criteria:

1. Patients currently taking hydroxychloroquine or related antimalarial such as mepacrine or chloroquine.
2. Patients with an estimated glomerular filtration rate (eGFR) <30 ml/min.
3. Patients weighing <40kg.
4. Sensitivity, anaphylaxis or allergy to hydroxychloroquine or any other 4-aminoquinoline compound.
5. Known glucose 6 phosphate dehydrogenase deficiency.
6. Known lactose intolerance.
7. Evidence of plaque psoriasis.
8. Concomitant use of the following medications within the last six months:

   Tumour necrosis factor inhibitor treatment (e.g. etanercept) Cyclophosphamide Abatacept Alemtuzumab Any experimental biological therapies Intravenous, intramuscular or sub-cutaneous immunoglobin Plasma exchange Antithymocyte globulin Tamoxifen Live vaccines
9. B cell depleting therapy (rituximab) for remission induction within the last six months. Rituximab maintenance therapy is permitted.
10. Severe or rapidly progressive ANCA vasculitis with at least one major BVAS item.
11. Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to vasculitis (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious disease) which, in the opinion of the principal investigator, could confound the results of the study or put the patient at undue risk.
12. Patients taking long term macrolide antibiotics for a chronic condition. This does not include topical preparations.
13. Have a history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
14. Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to randomisation. A urine drug screen should be performed and confirmed negative prior to study entry.
15. Have a historically positive test or test positive at screening for hepatitis B surface antigen, hepatitis B core antibody or hepatitis C antibody or are known to be HIV-1 positive.
16. Have a Grade 3 or greater laboratory abnormality based on the Common Terminology Criteria for Adverse Events (CTCAE) toxicity scale (version 5), unless considered by the investigator to be related to the underlying disease or induction therapy.
17. Screening 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect patient safety or interpretation of study results, including: - QT interval corrected using the same consistent formula at each visit (QTc) > 470 msec for female > 450 msec for male patients demonstrated by at least two ECGs.
18. Participation in any other interventional trial within the last 6 months.
19. Have a current symptomatic COVID-19 infection.
20. Have been admitted to the ICU in the past 6 months due to a COVID-19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with • uncontrolled AAV disease activity OR • controlled AAV disease activity but prednisolone dose >7.5mg daily OR • controlled AAV disease activity but any corticosteroid use >7.5mg daily for any reason | BVAS will be assessed during the final 12 (±7 days) weeks that the patient is on the study drug in the trial.
  The primary endpoint will be the percentage of patients with:
  EITHER
  * uncontrolled AAV disease activity (defined as BVAS > 3) OR
  * controlled AAV disease activity (BVAS ≤ 3) but prednisolone dose >7.5mg daily OR
  * controlled AAV disease activity (BVAS ≤ 3) but any corticosteroid use >7.5mg daily for any reason
  at any point during the final 12 weeks (±7 days) of the study.
  Inhaled corticosteroids will not contribute to the primary endpoint, nor will methylprednisolone given for rituximab maintenance therapy.

SECONDARY OUTCOMES:
Cumulative number of visits BVAS = 0 | Week 4 through to week 52
  Excluding screening, baseline and week 56
Proportion of patients with treatment failure at week 52 | Week 52
  As above
Cumulative prednisolone dosage | From date of randomisation through to week 56 follow up
  As above
Total number of adverse events | From date of randomisation through to week 56 follow up
  As above
Total number of infections per patient | From date of randomisation through to week 56 follow up
  As above
Total number of vasculitis flares (severe and limited) per patient | From date of randomisation through to week 56 follow up
  As above
Time to remission | From date of randomisation through to week 56 follow up
  As above
Time to first severe flare | From date of randomisation through to week 56 follow up
  Patients will be categorized as having a severe flare if they have a new or worsening major item on the BVAS.
  Proportion of patients with a limited disease flare defined as having a new or worsening minor BVAS item with no major items at each time point outlined in the trial flowchart.
Time to first limited flare | From date of randomisation through to week 56 follow up
  Patients will be categorized as having a limited flare if they have a new or worsening minor item on the BVAS with no new major items.
Proportion of patients categorized as having a severe flare at each of the time points in the trial schedule excluding screening, baseline and week 56 | Weeks 1-52 excluding screening, baseline and week 56
  As above
Proportion of patients categorized as having a limited flare at each of the time points in the trial schedule excluding screening, baseline and week 56 | Weeks 1-52 excluding screening, baseline and week 56
  As above
Absolute values and relative change from baseline in the Vasculitis Damage Index (VDI) at each time point outlined in the trial schedule. | From date of randomisation through to week 56 follow up
  As above

CONTACTS AND LOCATIONS:
Overall Officials: David D'Cruz, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (18):
- United Kingdom (18):
  - Royal Berkshire NHS Foundation Trust, Reading, Berkshire
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire
  - NHS Highland, Inverness, Inverness-shire
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside
  - Royal United Hospitals Bath NHS Foundation Trust, Bath, Somerset
  - Surrey and Sussex Healthcare NHS Trust, Redhill, Surrey
  - University Hospitals Sussex NHS Foundation Trust, Brighton, Sussex
  - Cardiff & Vale University Health Board, Cardiff
  - Epsom and St Helier University Hospitals NHS Trust, Epsom
  - Cwm Taf Morgannwg University Health Board, Llantrisant
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland
  - Torbay and South Devon NHS Foundation Trust, Torquay

IPD SHARING:
Plan to Share IPD: No
N/A - no plan to share identifiable patient data with other researchers.

REFERENCES:
- [Derived] Learoyd AE, Arnold L, Reid F, Beckley-Hoelscher N, Casian A, Sangle S, Morton N, Nel L, Cape A, John S, Kim S, Shivapatham D, Luqmani R, Jayne D, Galloway J, Douiri A, D'Cruz D; HAVEN study group. The HAVEN study-hydroxychloroquine in ANCA vasculitis evaluation-a multicentre, randomised, double-blind, placebo-controlled trial: study protocol and statistical analysis plan. Trials. 2023 Apr 6;24(1):261. doi: 10.1186/s13063-023-07108-3. PMID 37024906